CLINICAL TRIAL: NCT03357692
Title: Ultrasonic Preparation of the Implant Site in the All-on-Four Technique With Trans-sinus Implants
Brief Title: All-on-Four Implants With Ultrasonic
Acronym: Nobelsinus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enough patients have been enrolled
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the International Piezosurgery Academy, International Piezosurgery Academy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nobelsinus
Record Dates: First submitted 2017-11-23; First posted 2017-11-30 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Bone Atrophy, Alveolar
Keywords: all on four; piezoelectric; implant; trans-sinusal
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maxillary total edentulism (Experimental): all on four implant rehabilitation with trans-sinusal implants
  Interventions: Procedure: all on four implant rehabilitation

INTERVENTIONS:
Procedure: all on four implant rehabilitation — implant insertion after piezoelectric site preparation for trans-sinusal implants

SUMMARY:
The objective of this observational study is the radiographic evaluation of marginal bone remodeling after surgical implant insertion in an immediate loading all-on-four technique with trans-sinusal titanium implants, correlating the gingival thickness and the height of the implant prosthetic stump with the proportion of the abovementioned marginal bone remodeling.

DETAILED DESCRIPTION:
The extent of marginal bone remodeling around the neck of dental implants has been used for many years as a criterion for defining its long-term success.

In fact, the etiology of this Marginal Bone Loss has not yet been well understood, although many theories have been proposed to explain it.

The influence of the thickness of the mucous membrane on marginal bone loss was discussed elsewhere which suggests a protective action for the underlying soft tissue that recreates a kind of "biological amplitude" around the implant. Some studies have suggested that a marginally oscillating bone loss between 1.5 and 2.0 mm provides the vertical space for proper restoration of the biological amplitude. Some authors. published a study that demonstrated that, in crestal systems with switching platforms, a vertical thickness of soft tissue greater than 2 mm is effective in preventing periimplant crestal bone loss. However, the severity of the sample examined precludes the possibility of making definitive conclusions.

Recently other authors have shown significant marginal bone loss around implants with lower prosthetic implants than those with higher prosthetic prostheses, without however measuring the thickness of soft tissues and evaluating their influence. In particular, the extent of bone loss was extremely limited when the height of the stump was equal to or greater than 2 mm. From a theoretical point of view, a prosthetic abutment of at least 2 mm high, calculated from the apical margin of the crown to the platform of the implant, should provide adequate space for restoring the biological amplitude.

It can therefore be hypothesized that these two factors (the vertical thickness of soft tissues and the height of the prosthetic stump) are the expression of the same principle: the restoration of the biological amplitude around the implant's neck. From a clinical point of view it will be useful to determine which of the two factors is most important in preventing and limiting periimplant bone loss.

ELIGIBILITY:
Inclusion Criteria:

1. indications for implant insertion into the maxillary upper jaw, based on a careful diagnosis and treatment plan;
2. presence of a residual bone crest with a minimum surgical height of 4 mm at the maxillary sinus (bilaterally), and a thickness of at least 6 mm at the two distally programmed implant sites;
3. presence of a residual bone crest with a minimum surgical height of 10 mm at the anterior maxilla, and a thickness of at least 6 mm at the mesially programmed implant sites;
4. the bone crest should be healed (at least 6 months after the loss / extraction of the corresponding dental element);
5. no regenerated bone;
6. Plaque index below 25% and bleeding index less than 20%;
7. the buccal length of the adherent gingiva ≥ 4 mm;
8. age of the patient> 18 years;
9. systemic condition of the compensated patient (American Society of Anesthesiologist score < 2);

8) Patients should be able to examine and understand the protocol of study; 9) subscribing to informed consent.

Exclusion Criteria:

1. not treated diabetes
2. cardiovascular disease
3. incapability of maintaining a good oral hygiene

Min Age: 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
survival rate | two years after surgery
  percentage of implants surviving in oral cavity

SECONDARY OUTCOMES:
radiographic distance between crestal bone and implant platform | two years after surgery
  radiographically assessed

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr, Study Director — International Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malo P, Rangert B, Nobre M. "All-on-Four" immediate-function concept with Branemark System implants for completely edentulous mandibles: a retrospective clinical study. Clin Implant Dent Relat Res. 2003;5 Suppl 1:2-9. doi: 10.1111/j.1708-8208.2003.tb00010.x. PMID 12691645
- [Background] Agliardi EL, Tete S, Romeo D, Malchiodi L, Gherlone E. Immediate function of partial fixed rehabilitation with axial and tilted implants having intrasinus insertion. J Craniofac Surg. 2014 May;25(3):851-5. doi: 10.1097/SCS.0000000000000959. PMID 24820712